CLINICAL TRIAL: NCT06896838
Title: Comparison of Intercostal and Quadriceps Femoris Muscle Oxygenation During Upper Extremity and Lower Extremity Maximal Exercise Tests in Women and Men
Brief Title: Comparison of Intercostal and Quadriceps Femoris Muscle Oxygenation in Women and Men
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Başak KAVALCI KOL, Principle Investigator, Kirsehir Ahi Evran Universitesi
Other Study IDs: AhiEvranU528
Record Dates: First submitted 2025-03-10; First posted 2025-03-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Near-Infrared Spectroscopy
Keywords: muscle oxygenation; exercise capacity; body composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female Group: Healthy, active individuals with no history of respiratory, cardiovascular, metabolic, musculoskeletal or acute infection at least 2 weeks before the test will be included in the study. Individuals whose activity level is in category 3 according to the International Physical Activity Questionnaire results (at least 3 days of vigorous activity providing a minimum of 1500 metabolic equivalent (MET)-minutes (min)/week or more days of walking, moderate or vigorous activity providing a minimum of 3000 MET-min/week, 7 or more days) will be included.
- Male Group: Healthy, active individuals with no history of respiratory, cardiovascular, metabolic, musculoskeletal or acute infection at least 2 weeks before the test will be included in the study. Individuals whose activity level is in category 3 according to the International Physical Activity Questionnaire results (at least 3 days of vigorous activity providing a minimum of 1500 MET-min/week or more days of walking, moderate or vigorous activity providing a minimum of 3000 MET-min/week, 7 or more days) will be included.

SUMMARY:
The differences in physiological responses due to gender during exercise tests have recently begun to be investigated. The oxygen use of respiratory muscles and lower extremity muscles may differ during upper and lower extremity exercise tests, but there is no study on this subject in the literature. The primary aim of this study was to compare intercostal and quadriceps femoris muscle oxygenation during upper extremity and lower extremity maximal exercise tests in women and men. The secondary aim of the study was to investigate the relationship between intercostal and quadriceps femoris muscle oxygenation and upper extremity and lower extremity exercise capacity, body composition, respiratory muscle strength, and respiratory muscle endurance in women and men.

DETAILED DESCRIPTION:
Differences in physiological responses due to gender during exercise tests have recently been investigated. In a study, it was determined that respiratory muscles such as intercostals use more oxygen during exercise tests in women. It was shown that this situation is related to the smaller rib cage, mechanical disadvantage of the diaphragm, narrower airway diameter and greater activation of accessory respiratory muscles in women. The fact that respiratory muscles consume more oxygen in women causes blood flow to the respiratory muscles to be higher. This situation causes a decrease in the amount of oxygen carried to the peripheral muscles, which may cause early fatigue in the peripheral muscles during the exercise test. Muscle oxygen saturation (SmO2) indicates the oxygen uptake and oxygen consumption of the muscle. This can be determined using continuous wave near infrared spectroscopy (NIRS, 630-850 nm) device, which measures changes in the amount of hemoglobin bound to oxygen at the microvascular level. Research on gender-related differences and how SmO2 levels in these muscles change during exercise in women is limited. The aim of the study was to compare intercostal and quadriceps femoris muscle oxygenation during upper extremity and lower extremity maximal exercise tests in women and men.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years,
* Physically active (doing moderate intensity physical activity 3 days a week for 150 minutes / week)
* Volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Healthy individuals with any diagnosed chronic or systemic disease,
* Those who smoke 10 packs x years or more,
* Those with pneumonia or any acute infection,
* Those with any psychiatric disorder will not be included in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Active individuals who are healthy, with no history of respiratory, cardiovascular, metabolic, musculoskeletal, or acute infections for at least 2 weeks prior to testing will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Maximal symptom limited cycle ergometer test | First day
  In order to evaluate the exercise capacity of individuals, a symptom-limited increasing workload exercise test will be applied on a bicycle ergometer. In the test, patients will warm up at 0 watts for 3 minutes and then proceed to the loading period of the test. During the loading period, patients will be provided with a 20-watt workload increase every 2 minutes to reach their maximal workload. Patients will be encouraged to continue testing to the maximum level they can sustain during the test. The test will be terminated by the practitioner when patients reach their maximal heart rate or if they wish to terminate the test due to symptoms.
Maximal symptom limited arm ergometer test | Second day
  Arm ergometer test will be used to evaluate the upper extremity exercise capacity of individuals. The test will be performed in a sitting position with the ergometer height at shoulder level. The arm ergometer test will begin at 0 watts (W) workload and 45-55 rpm at each stage. The workload will be increased by 10 W every two minutes. The highest workload reached during the test will be recorded as watt.
Evaluation of Quadriceps Femoris Muscle Oxygenation | First day
  Muscle oxygen level and total hemoglobin level of quadriceps femoris will be measured using Moxy® monitor (Moxy, Fortiori Design LLC, Minnesota, USA) before cycle ergometer test, during testing and during post-test recovery.
Evaluation of Intercostals Muscle Oxygenation | Second day
  Muscle oxygen level and total hemoglobin level of and intercostal muscles will be measured using Moxy® monitor (Moxy, Fortiori Design LLC, Minnesota, USA) before arm ergometer test, during testing and during post-test recovery.

SECONDARY OUTCOMES:
Evaluation of respiratory muscle strength | Second day
  n the evaluation of respiratory muscle strength, an electronic mouth pressure device will be used, which complies with American Thoracic Society and European Respiratory Society criteria. Maximal inspiratory pressure and maximal expiratory pressures of the individuals will be measured with the mouth pressure measuring device.
Evaluation of respiratory muscle endurance | Second day
  The incremental threshold workload test will be used to evaluate respiratory muscle endurance. The PowerBreathe Wellness® (HaB International Ltd. Southam, UK) inspiratory muscle trainer will be used in the incremental threshold load test. The measurement will start with 30% of the maximal inspiratory pressure. Every two minutes, pressures will be increased by 10%. At the end of the test, the highest pressure value that the participants can maintain for one minute will be recorded in centimetre of water pressure and the total time will be recorded in seconds, and the respiratory muscle endurance result value will be calculated by multiplying these two result values
Evaluation of body composition | First day
  Total body weight, body fat percentage and body fat percentage of individuals will be evaluated by bioelectrical impedance analysis system. Bioelectrical impedance analyzer is a high-speed, low-cost and non-invasive device. The device provides low-dose and different-frequency electrical current to the body. Impedance analysis expresses the resistance of body tissues to this low-dose electrical transmission and is inversely proportional to conductivity. While bone and fat tissue encounter stronger resistance during different electrical current advances, muscle tissue and visceral organs encounter lower resistance during transmission. In this way, it provides information about body fat, bone and muscle ratios. The device will thus present data such as body fat percentage and body fat ratio as output in a single report with the different electrical currents it sends. Bioelectrical impedance analysis measurements have a good level of reliability (ICC≥0.82).

CONTACTS AND LOCATIONS:
Overall Officials: Başak KAVALCI KOL, PhD, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Physical Therapy and Rehabilitation Center, Cardiopulmonary Unit, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In the study, all data will be stored in a locked cabinet.